CLINICAL TRIAL: NCT07066774
Title: Diagnostic Accuracy of Different Tru-Cut Needle Sizes in Soft Tissue Sarcomas: A Prospective Blinded Study
Brief Title: Biopsy Needle Size in Soft Tissue Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Geotek Medical Products Industry and Trade Co., Ltd., Ankara, Türkiye (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: E2-25-10025
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Soft Tissue Sarcoma of the Limb
Keywords: needle size, soft tissue sarcoma, diagnostic accuracy
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 14G Needle (Experimental): Each patient undergoes a tru-cut biopsy with a 14 G needle, obtaining 5 tissue cores (tumor center, superior, inferior, medial, lateral).
  Interventions: Diagnostic Test: Tru-cut Biopsy with 14 G Needle
- 16G Needle (Experimental): Each participant underwent Percutaneous Tru-cut Biopsy with 16G tru-cut needles in a single session procedure and within-subject repeated measuring data is obtained
  Interventions: Diagnostic Test: Tru-cut Biopsy with 16G tru-cut needle
- 18G Needle (Experimental): Each participant underwent Percutaneous Tru-cut Biopsy with 16G tru-cut needles in a single session procedure and within-subject repeated measuring data is obtained
  Interventions: Diagnostic Test: Tru-cut Biopsy with 18G tru-cut needle

INTERVENTIONS:
Diagnostic Test: Tru-cut Biopsy with 14 G Needle — Each participant underwent Percutaneous Tru-cut Biopsy with 14G tru-cut needle in a single session procedure. There are no studies to our knowledge to compare samples from the same tumor
  Arms: 14G Needle
Diagnostic Test: Tru-cut Biopsy with 16G tru-cut needle — Each participant underwent Percutaneous Tru-cut Biopsy with 16 tru-cut needle in a single session procedure. There are no studies to our knowledge to compare samples from the same tumor
  Arms: 16G Needle
Diagnostic Test: Tru-cut Biopsy with 18G tru-cut needle — Each participant underwent Percutaneous Tru-cut Biopsy with 18G tru-cut needle in a single session procedure. There are no studies to our knowledge to compare samples from the same tumor
  Arms: 18G Needle

SUMMARY:
Soft tissue sarcomas (STS) require accurate biopsy for diagnosis, grading, and management decisions. Although tru-cut biopsy is widely used, the optimal needle gauge remains uncertain. This study aimed to compare diagnostic accuracy and biopsy concordance rates of 14 G, 16 G, and 18 G tru-cut biopsy needles for extremity STS.

1. Is there any difference between the diagnostic accuracy measurements of 14G, 16G and 18G tru-cut biopsy needles for diagnosis of soft tissue sarcomas in extremities?
2. Do tumor size, tumor depth, tumor subtype and histological grade of the tumor affect the "matching score"s of biopsies?
3. Do tumor size, tumor depth, tumor subtype and histological grade of the tumor affect the biopsy result concordance and/or diagnostic accuracy measurements?
4. Does needle gauge effect successful tumoral tissue sampling or prediction of histological grade of soft tissue sarcomas?

DETAILED DESCRIPTION:
In 2018, the National Comprehensive Cancer Network (NCCN) endorsed core-needle (tru-cut) biopsy as the preferred diagnostic modality for STSs [14]. They recommend obtaining at least three tissue core blocks through a single stab incision on the skin, with a 14-gauge needle, directing the needle along different trajectories. In clinical practice, both 14 G and 16 G cores are commonly used Although multiple tru-cut needle gauges are used in practice, to our knowledge, an ideal and safe biopsy needle that does not sacrife diagnostic performance has not been defined. This is a randomized prospective disagnostic accuracy study. Therefore we prospectively compared numerous variables (tumor size, tumor depth, subtype, histological grade etc.) with biopsy result concordance and diagnostic accuracy of 14 G, 16 G, and 18 G tru-cut needles in samples obtained from the same tumor for each patient with suspected extremity STS, to determine whether an optimal needle gauge exists.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Orthopedic Oncology outpatient clinic at Ankara Bilkent City Hospital with suspected or preliminary findings on physical examination suggesting soft tissue sarcoma.

Patients presenting to the Orthopedic Oncology outpatient clinic at Ankara Bilkent City Hospital with suspected or preliminary findings on radiological imaging suggesting soft tissue sarcoma.

Patients with soft tissue masses in extremities which require pathological examination

Exclusion Criteria:

* Patients with a prior diagnosis of the existing mass, coagulation disorders, active infection at the tumor site, a history of previous surgery or radiotherapy to the tumor region, medical conditions contraindicating tru-cut biopsy, or those who did not consent to participate after detailed explanation of the study, were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy methods | From enrollment to the end of study at 4 months
  Sensitivity, specificity, positive predictive value, negative predictive value, false positive rate and false negative rate was analyzed for 3 different needle sizes

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will no affect the study results or analysis.

REFERENCES:
- [Background] Birgin E, Yang C, Hetjens S, Reissfelder C, Hohenberger P, Rahbari NN. Core needle biopsy versus incisional biopsy for differentiation of soft-tissue sarcomas: A systematic review and meta-analysis. Cancer. 2020 Jan 1;126(9):1917-1928. doi: 10.1002/cncr.32735. Epub 2020 Feb 5. PMID 32022262